CLINICAL TRIAL: NCT02150720
Title: Prevention of Postoperative Bleeding in Femoral Fractures: a Multicenter, Randomized, Controlled, Parallel Clinical Trial to Assess the Efficacy of Tranexamic Acid and Fibrin Glue
Brief Title: Prevention of Postoperative Bleeding in Subcapital Femoral Fractures
Acronym: TRANEXFER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-FAT-2011-103; EC11-341 (Other Grant/Funding Number: Ministry of Health and Social Policy 2011); 2011-006278-15 (EudraCT Number); SA/12/AYU/456 (Other Grant/Funding Number: Fundación MAPFRE 2012)
Record Dates: First submitted 2014-05-22; First posted 2014-05-30 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Hip Fracture; Blood Loss
Keywords: Hip fractures; Clinical Trial; Randomized; Fibrin glue; Tranexamic acid; Blood loss
MeSH Terms: conditions — Hip Fractures; Hemorrhage | interventions — Tranexamic Acid; Fibrin Tissue Adhesive; Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tranexamic acid (Experimental): Tranexamic acid, 1g intra-articular before closing the surgery wound
  Interventions: Drug: Tranexamic Acid; Procedure: Electrocauterization
- Fibrin glue (Experimental): One intra-articular dose of fibrin glue (Evicel 5mL) before closing the wound surgery,
  Interventions: Drug: Fibrin glue; Procedure: Electrocauterization
- Usual hemostasia (Active Comparator): Electrocauterization
  Interventions: Procedure: Electrocauterization

INTERVENTIONS:
Drug: Tranexamic Acid — 1g intra-articular before closing the wound surgery
  Other Names: Amchafibrin
  Arms: Tranexamic acid
Drug: Fibrin glue — 5mL intra-articular before closing the wound surgery
  Other Names: Evicel
  Arms: Fibrin glue
Procedure: Electrocauterization — Coagulation blood from vessels by means of a electrocautery.

SUMMARY:
The main hypothesis of this clinical trial is that the use of intra-articular tranexamic acid and the fibrin glue plus usual hemostasis will reduce at least a 25% the postoperative blood loss with respect to usual hemostasis in patients undergoing subcapital femoral fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patients with unilateral subcapital femoral fracture
* Patients requiring hip replacement (total or partial)
* Signed informed consent from the patient or legal representative

Exclusion Criteria:

* Known allergy to fibrin glue and tranexamic acid
* Multiple fractures
* Pathological fractures
* Contraceptives or estrogen therapy
* Use of blood salvage during surgery
* History compatible with thromboembolic disease:

  * Cerebral vascular accident
  * Ischemic heart disease (myocardial infarction, angina )
  * Deep vein thrombosis
  * Pulmonary Embolism
  * Peripheral arterial vasculopathy
  * Patients with thrombogenic arrhythmias
  * Patients with cardiovascular stents
  * Prothrombotic alterations in coagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2013-02; Primary Completion 2015-04 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Blood loss (ml) after surgery | The first postoperative 24h
  The blood lost from the wound will be collected by a drainage system during the first 24 hours postoperatively.

SECONDARY OUTCOMES:
Hidden blood loss | The first postoperative five days
  The hidden blood loss is the total blood loss calculated by the formula of Nadler minus the blood loss by drain.
Proportion of patients requiring blood transfusion | The first postoperative ten days
Units of blood transfused | The first postoperative ten days
Proportion of patients with wound infection | The first postoperative month
Proportion of patients with wound dehiscence | The first postoperative month
Deep venous thrombosis | The first postoperative ten days
Length of hospital stay | The first postoperative ten days
  Time from hip surgery until hospital discharge
Quality of life measured with the generic EQ-5D -5L | Preoperatively, at 5 days postoperatively , 1-2, 6 and 12 months postoperative follow-up
Mortality | During the 12 month of follow-up after surgery
Direct cost | During the first postoperative month

CONTACTS AND LOCATIONS:
Overall Officials: MJ Martínez-Zapata, MD, PhD, Principal Investigator — Iberoamerican Cochrane Centre. Research Institut Hospital de la Santa Creu i Sant Pau. IIB Sant Pau
Locations (6):
- Spain (6):
  - Hospital Germans Trias i Pujol de Badalona, Badalona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Clinic, Barcelona, Barcelona
  - Parc Taulí, Sabadell, Barcelona
  - Hospital Universitari Mútua Terrassa, Terrassa, Barcelona
  - Hospital Universitari Terrassa-Consorci Sanitari de Terrassa, Terrassa, Barcelona

REFERENCES:
- [Result] Martínez-Zapata MJ, Jordán M, Aguilera X, Cánovas E, Urrutia G (en nombre del grupo TRANEXFER). Estudio prospectivo multicéntrico de una cohorte para evaluar la calidad de vida de pacientes intervenidos de fractura subcapital de fémur. Trauma 2014; 25 (4): 188-195.
- [Derived] Merchan-Galvis A, Posso M, Canovas E, Jordan M, Aguilera X, Martinez-Zapata MJ. Quality of life and cost-effectiveness analysis of topical tranexamic acid and fibrin glue in femur fracture surgery. BMC Musculoskelet Disord. 2022 Aug 31;23(1):827. doi: 10.1186/s12891-022-05775-y. PMID 36045358
- See also: Publication of quality of life (subgroup of patients) — http://www.mapfre.com/fundacion/html/revistas/trauma/v25n4/docs/v25n4.pdf